CLINICAL TRIAL: NCT03273738
Title: Assessment of Vascular and Metabolic Changes in Post-menopausal Women With Type 2 Diabetes Mellitus
Brief Title: Vascular and Metabolic Changes in Postmenopausal Diabetics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed, principal investigator, Assiut University
Other Study IDs: Postmenopausal DM
Record Dates: First submitted 2017-08-30; First posted 2017-09-06 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Diabete Type 2
Keywords: type 2 diabetes; postmenopausal
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postmenopausal diabetic women: 50 female patients with T2DM who visited Assiut University Hospital Diabetes Clinic in Assiut, Egypt in these patients folate level measurement, B12 level and homocysteine are measured
  Interventions: Diagnostic Test: folate level measurement; Diagnostic Test: B12
- postmenopausal without diabetes: Another 50 participants will be volunteered in the study as control.n these subjects folate level measurement', B12 level and homocysteine are measured
  Interventions: Diagnostic Test: folate level measurement; Diagnostic Test: B12

INTERVENTIONS:
Diagnostic Test: folate level measurement — the level of folate measured in plasma with homocysteine
Diagnostic Test: B12 — B12 measurement in blood

SUMMARY:
The presence of type 2 diabetes mellitus (T2DM) also increases the relative risk of developing cardiovascular disease in women compared to men. Carotid intima media thickness (IMTc) was increased with reduction in brachial artery flow-mediated dilation (FMD) in T2 DM patients and inversely and strongly related to the extent of hyperglycemia. Low concentrations of folate and vitamin B12 involved in homocysteine metabolism are also associated with increased risk of vascular damage. the aim is to relate, if found, the degree of metabolic changes to the extent in vascular parameters changes in type 2 diabetic postmenopausal women.

DETAILED DESCRIPTION:
Introduction Complications of diabetes, such as cardiovascular disease, are associated with increased mortality among type 2 diabetes mellitus patients. The presence of type 2 diabetes mellitus (T2DM) also increases the relative risk of developing cardiovascular disease in women compared to men . Major cardiovascular disease risk factors that have been identified in T2DM patients include arterial stiffening, endothelial dysfunction, hyperglycemia , and elevated glycated haemoglobin (HbA1c) concentrations.

Cardiovascular disease is the major cause of morbidity and mortality in T2 DM, due to arterial structure and functional changes. Evaluation of vascular dysfunction in T2 DM patients include: carotid intima media thickness (IMTc), pulse wave velocity (PWV), and brachial artery flow-mediated dilation (FMD). IMTc is increased in patients with T2 DM with reductions in FMD, which have already been reported to be inversely and strongly related to the extent of hyperglycemia.

The incidence of vascular complications is multifactorial and may not be explained by hyperglycemia alone. Other presumably unrelated risk factors, such as hyperhomocysteinemia may be involved in the atherothrombotic process. High levels of homocysteine have been identified as a risk factor for cardiovascular disease in T2DM patients. Levels of plasma homocysteine increase in women after menopause, and postmenopausal diabetic women are consequently at significantly increased risk of cardiovascular disease.

High concentrations of homocysteine are associated with increased low-density lipoprotein oxidation, endothelial dysfunction, dysfunction of β-islet cells and inhibiting secretion of insulin. Also, hyperhomocysteinemia was an independent risk factor for the occurrence of diabetic peripheral neuropathy .

In newly diagnosed normotensive T2DM patients, the left ventricular mass index (LVMI), carotid intima media thickness (CIMT), and creatinine levels and 24-hr microalbuminuria were used to determine cardiac, carotid, and kidney end-organ diseases, respectively. It was found that, LVMI, CIMT, and creatinine level were positively correlated with the homocysteine level.

Moreover, determinants of hyperhomocysteinemia, such as low concentrations of folate and vitamin B12 involved in homocysteine metabolism are also associated with increased risk of vascular damage. Folic acid supplementation may improve the cardiovascular health of post-menopausal women with diabetes, reduce homocysteine levels and improve vascular health in different study populations.

Increased plasma homocysteine, triglyceride and waist circumference as well as decreased folic acid and vitamin B12 in type 2 diabetes mellitus were evaluated.

Sudchada et al. concluded that folic acid supplementation in patient with T2DM may reduce total homocysteine levels and have a trend to associate with better glycemic control compared with placebo.

in postmenopausal Korean women with type 2 diabetes mellitus, folic acid supplementation reduced serum homocysteine levels, increased serum folate and vitamin B12 levels, and lowered lipid parameters.

A case-control study showed that low intakes of folate and B12 in type 2 diabetic patients were associated with hyperhomocysteinemia. Additionally, folate has also been shown to improve glycemic control by reducing glycosylated hemoglobin fasting blood glucose, serum insulin and insulin resistance as well as homocysteinemia in type 2 diabetes patients.

Folic acid supplementation significantly reduced LDL-C levels as well as LDL-C/HDL-C and TC/HDL-C ratios. The improvements in lipid parameters might be due to the reduction of serum homocysteine levels caused by folic acid supplementation. In another study, associations between fasting plasma homocysteine concentration and age, serum creatinine, and vitamin B12. However, no association between folate and homocysteine was found.

Whether serum homocysteine levels are associated with coronary heart disease (CHD) and the metabolic syndrome (MS) needs investigation in different ethnic groups. High serum homocysteine and low folate levels are associated in Turkish men independently with coronary heart disease, which needs confirmation in a larger sample. In women, vitamin B12 concentrations are significantly associated with metabolic syndrome likelihood.

there is no support that metformin consumption increases homocysteine secondary to folate and /or B12 deficiency in patients with T2DM. Also, among adults with hypertension with no history of stroke and/or myocardial infarction, folic acid supplementation had no significant effect on the risk of new-onset diabetes.

However, clinical studies have shown that folic acid therapy is not very effective in normalizing hyperhomocysteinemia in uremic patients. Indeed, it has been demonstrated that vitamin B12 supplementation alone, or in combination with folic acid, decreases total homocysteine concentrations, but full normalization is not achieved. folate levels were comparable to controls at various chronic kidney disease stages, whereas vitamin B12 levels were lower, except at stage IV in patients with T2DM. They did not find any correlation between B-vitamins and levels of total homocysteine and cysteine, regardless of the CKD stage.

Aims of the study:

1. To evaluate cardiovascular changes in type 2 diabetic postmenopausal women through measurement of vascular parameters.
2. To assess the possible changes in some metabolic features in type 2 diabetic postmenopausal women.
3. To relate, if found, the degree of metabolic changes to the extent in vascular parameters changes in type 2 diabetic postmenopausal women.

Type of study and its design:

Study subjects:

This study will include 50 female patients with T2DM who visited Assiut University Hospital Diabetes Clinic in Assiut, Egypt. Another 50 participants will be volunteered in the study as control.

Inclusion criteria:

For this study, 100 post-menopausal women aged 50-70 years with amenorrhea for over 24 months will be recruited. The diabetic participants will receive their treatment for T2DM (oral hypoglycemic agents or insulin).

Exclusion criteria:

1. Patients receiving hormone replacement therapy.
2. History of abnormal vaginal bleeding.
3. Patients receiving vitamin B12, vitamin D and folic acid regularly.
4. History of malignancy or neurological diseases as epilepsy, parkinsonism and Alzheimer disease.
5. Antifolate medications as methotrexate are excluded from the study.

Study design:

The study will be observational study. The participants will be informed about the study and we will take their assignment on written consent. The patients included will be divided into two groups. 20 healthy participants and 100 female patients, will be subjected to clinical evaluation and blood sampling for laboratory investigations.

Evaluation of the patients:

All patients will be subjected to:

1. Complete history (age, occupation, menstrual history, bleeding tendency, renal disease, therapeutic and dietary history)
2. Clinical examination (weight, height, blood pressure measurement, presence of microvascular or macrovascular complications, anemia).
3. ECG.
4. Brachial-ankle pulse wave velocity (baPWV) will be calculated further using the following equation:

   baPWV = transmission distance/transmission time
5. Carotid intima-media thickness (CIMT) will be done, it is noninvasive measure that uses ultrasound to detect the presence and extent of atherosclerosis.
6. Laboratory investigations:

   1. HbA1c.
   2. Lipid profiles (total cholesterol, LDL-C, HDL-C and triglycerides)
   3. Serum homocysteine will be measured using available commercial ELISA kits.
   4. Serum folic acid level will be measured using available commercial ELISA kits.

   <!-- -->

   1. Serum vitamin B12 level will be measured using available commercial ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women
* aged 50-70 years
* amenorrhea for over 24 months.
* The diabetic participants will receive their treatment for T2DM (oral hypoglycemic agents or insulin).

Exclusion Criteria:

* Patients receiving hormone replacement therapy.
* History of abnormal vaginal bleeding.
* Patients receiving vitamin B12, vitamin D and folic acid regularly.
* History of malignancy or neurological diseases as epilepsy, parkinsonism and Alzheimer disease.
* Antifolate medications as methotrexate are excluded from the study.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Study Population: post-menopausal women aged 50-70 years with amenorrhea for over 24 months will be recruited. The diabetic participants will receive their treatment for T2DM (oral hypoglycemic agents or insulin).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-02 (Estimated); Primary Completion 2018-10-10 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
metabolic changes in type 2 diabetes | baseline and 3 months
  changes in folate level in type 2 diabetes mellitus
metabolic changes in type 2 diabetes | baseline and 3 months
  B12 level and their relation to complications

CONTACTS AND LOCATIONS:
Overall Officials: Lobna F Eltoony, Study Chair — internal medicine

IPD SHARING:
Plan to Share IPD: Undecided
share measurements results in medical journals